CLINICAL TRIAL: NCT00592007
Title: Phase II Trial Evaluating Addition of Fulvestrant to Erlotinib in Patients With Stage IIIB/IV NSCLC Who Are Stable on Erlotinib and Exhibit Positivity for Estrogen or Progesterone Receptor
Brief Title: Study Evaluating the Addition of Fulvestrant to Erlotinib in Stage IIIB/IV Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to slow subject accrual
Sponsor: Lyudmila Bazhenova, M.D. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Lyudmila Bazhenova, M.D., Assistant Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD-060769; HRPP# 060769
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Non Small Cell Lung Cancer; Stage IIIB; Stage IV; Stable on Erlotinib; Exhibit Positivity for Estrogen or Progesterone Receptor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fulvestrant; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Single-arm study
  Interventions: Drug: Fulvestrant and Erlotinib

INTERVENTIONS:
Drug: Fulvestrant and Erlotinib — Upon enrollment, patients will continue to receive erlotinib daily orally at 150 mg/day or at 100 mg/day if 150 mg was associated with adverse events requiring dose reduction before enrollment in this study. Doses less than 100 mg/day will not be allowed. Fulvestrant will be added intramuscularly 500 mg Day 0, 250 mg Days 14 and 28. In cycles 2 and up, fulvestrant will be given 250 mg on day 28. Patients will receive this therapy until they progress.
  Other Names: Faslodex and Erlotinib

SUMMARY:
The main purpose of this research study is to see if adding fulvestrant (Faslodex) to erlotinib (Tarceva) is effective in patients with stage IIIb/IV Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
Erlotinib is an oral drug which is able to block endothelial growth factor receptor (EGFR). EGFR stimulates cancer cell growth. Fulvestrant (faslodex) block estrogen hormone from gaining access to tumor and stimulating the tumor cells to grow. Both of these drugs are already approved by FDA but have not been studied in this combination.

We will study if the combination of these drugs will delay treatment failure. Lung cancer tumors in both males and females can be sensitive to estrogen. Only patients whose tumor expresses the estrogen will be eligible for the trial. Estrogen sensitivity will be tested on previously removed tumor specimens.

ELIGIBILITY:
Inclusion Criteria:

* Estrogen or progesterone receptor positive stage IIIb/IV non-small cell lung cancer
* Eligible patients will have stable disease on erlotinib monotherapy at FDA- approved doses after a minimum duration of erlotinib therapy of 2 months
* 18 years or older
* ECOG Performance Status ≤2
* Adequate Organ Function Requirements
* Adequate coagulation function
* Postmenopausal status in female patients is required and is defined as no menstrual periods for 12 month or surgical menopause
* All patients must sign a written informed consent.

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study
* Patients who are currently receiving another investigational drugs
* Patients who are currently receiving other anti-cancer agents.
* Hormone replacement therapy will not be allowed and have to be stopped 1 month prior to entry into the study
* Patients who have an uncontrolled infection.
* Patients receiving less than 100mg/day of erlotinib
* Patients with evidence of progression after 2 months of erlotinib monotherapy.
* Patients with a history of bleeding diathesis (i.e., disseminated intravascular coagulation [DIC], clotting factor deficiency) or long-term anticoagulant therapy (other than antiplatelet therapy).
* Patients with a history of hypersensitivity to active or inactive excipients of fulvestrant (i.e. castor oil or Mannitol).
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-09; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyudmila Bazhenova, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

REFERENCES:
- See also: Moores UCSD Cancer Center Homepage — http://cancer.ucsd.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Fulvestrand and Erlotinib: Single-arm study
  Fulvestrant and Erlotinib : Upon enrollment, patients will continue to receive erlotinib daily orally at 150 mg/day or at 100 mg/day if 150 mg was associated with adverse events requiring dose reduction before enrollment in this study. Doses less than 100 mg/day will not be allowed. Fulvestrant will be added intramuscularly 500 mg Day 0, 250 mg Days 14 and 28. In cycles 2 and up, fulvestrant will be given 250 mg on day 28. Patients will receive this therapy until they progress.
Period: Overall Study
Arm/Group | Fulvestrand and Erlotinib
Started | 7
Completed | 5
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — patient ineligible (out of lab range) | 1

BASELINE CHARACTERISTICS:
Groups:
- Fulvestrant and Erlotinib: Single-arm study
  Fulvestrant and Erlotinib: Upon enrollment, patients will continue to receive erlotinib daily orally at 150 mg/day or at 100 mg/day if 150 mg was associated with adverse events requiring dose reduction before enrollment in this study. Doses less than 100 mg/day will not be allowed. Fulvestrant will be added intramuscularly 500 mg Day 0, 250 mg Days 14 and 28. In cycles 2 and up, fulvestrant will be given 250 mg on day 28. Patients will receive this therapy until they progress.
Arm/Group | Fulvestrant and Erlotinib
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Time Frame: 14 weeks after start of fulvestrant
Population: Subjects did not complete the study as planned. Zero participants analyzed due to termination of study. Data were not collected for this Outcome Measure. Outcomes were not collected due to withdrawal of the funding. Data not available.
Groups:
- Arm A: Single-arm study
  Fulvestrant and Erlotinib: Upon enrollment, patients will continue to receive erlotinib daily orally at 150 mg/day or at 100 mg/day if 150 mg was associated with adverse events requiring dose reduction before enrollment in this study. Doses less than 100 mg/day will not be allowed. Fulvestrant will be added intramuscularly 500 mg Day 0, 250 mg Days 14 and 28. In cycles 2 and up, fulvestrant will be given 250 mg on day 28. Patients will receive this therapy until they progress.
Arm/Group | Arm A
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Time Frame: Patients will be followed until death
Population: as for outcome 1
Arm/Group | Arm A
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- A: Fulvestrant and Erlotinib: Single-arm study
  Fulvestrant and Erlotinib: Upon enrollment, patients will continue to receive erlotinib daily orally at 150 mg/day or at 100 mg/day if 150 mg was associated with adverse events requiring dose reduction before enrollment in this study. Doses less than 100 mg/day will not be allowed. Fulvestrant will be added intramuscularly 500 mg Day 0, 250 mg Days 14 and 28. In cycles 2 and up, fulvestrant will be given 250 mg on day 28. Patients will receive this therapy until they progress.
Arm/Group | A: Fulvestrant and Erlotinib
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Fulvestrant and Erlotinib (N=7)
Acneiform Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology - Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Pain - Arthralgia (Nervous system disorders) | 1 (1)
Paronychia (Skin and subcutaneous tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Bronchorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash in Groin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Left Groin Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Changes in Equilibrium (Ear and labyrinth disorders) | 1 (1)
Double Vision (Nervous system disorders) | 2 (2)
Night Sweats (Immune system disorders) | 1 (1)
Hot Flashes (Endocrine disorders) | 3 (3)
Decreased Appetite (General disorders) | 1 (1)
Weight Loss (General disorders) | 2 (2)
Right Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Draining Sinuses (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Cardiac Murmur (Cardiac disorders) | 1 (1)
ALT Elevated (Investigations) | 1 (1)
AST Elevated (Investigations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: embargo of 60 days or less